CLINICAL TRIAL: NCT05167474
Title: Influence of Breast Milk Smell on Newborns Bilirubin Level, Duration of Time Phototherapy and Comfort in Newborns Receiving Phototherapy
Brief Title: Influence of Breast Milk Smell on Newborns Bilirubin Level, Duration of Time Phototherapy and Comfort in Newborns Receiving Phototherapyv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Elif Nilay Kizilay, nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: ENilayKizilay
Record Dates: First submitted 2021-11-10; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Newborn Jaundice
Keywords: newborn; phototherapy; breast milk smell
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breast milk smell (Active Comparator): The application of maternal education for the phototherapy method for newborns is to place the cotton unloaded by the mother in a container and place it close to the shape.
  Interventions: Other: breast milk smell
- control group (No Intervention): No intervention was performed during phototherapy treatment in newborns.

INTERVENTIONS:
Other: breast milk smell — yenidoğanlara fototerapi tedavisi esnasında anne sütü kokusu uygulanmıştır.
  Other Names: kontrol grubu
  Arms: breast milk smell

SUMMARY:
ABSTRACT Purpose: This research was done for the purpose of determining the impact of breast milk smell administered to term infants hospitalized in neonatal intensive care units (NICU) due to physiological jaundice on their bilirubin levels, length of remaining in phototherapy and comfort.

Material and Method: It is an experimental, randomisation, controlled research. Target population of the research consisted of a total of 72 term infants who were hospitalized in the NICU of Bilecik Bozuyuk Public Hospital and met the sample selection criteria. Our research includes two groups. Breast milk smell group and control group. The infants were assigned to the groups via randomization method. Sample assignment to the groups was performed using stratification and blocking methods. The infants meeting the research sample selection criteria were stratified according to their postnatal age and then assigned to each group equally (blocking) by lot. However, two infants in the control group were excluded from the research at the request of their parents as the research continued. Thus, the research was completed with a total of 72 infants; 37 in the breast milk smell group and 35 in the control group. In the research, the data were collected using "Personal Data Collection Form", "Phototherapy Follow-up Chart" and "Neonatal Comfort Behavior Scale". The data were analyzed using the SPSS (Statistical Package for Social Sciences) 21.0 (IBM corp. Relased 2012. IBM SPSS Statistics for Windows, version 21.0 Armonk, NY: IBM corp.) package software.

ELIGIBILITY:
Inclusion Criteria:

* The term baby (37-39+6 weeks) of the newborn according to the menstruation of the mothers
* Need to have phototherapy treatment for the first time
* Not taking analgesics and/or sedatives in the last 24 hours
* Body weight in the range of 2500 - 4000 g
* Postnatal age of the newborn greater than 48 hours
* Turkish Neonatology Society's approach, follow-up and treatment guideline for neonatal jaundice (2014) Being a medium and high risk baby according to the table of risk status determination of babies according to postnatal age and transcutaneous or total serum bilirubin values.
* Not taking any treatment or medication other than phototherapy treatment
* The mother and/or father accepting the study is having a baby.

Exclusion Criteria:

* Having a health problem other than physiological jaundice
* Findings such as tachypnea, fever
* Having an invasive procedure other than blood sampling once a day for babies
* Exchanged babies
* Babies with Rh and AB0 incompatibility
* Babies with elevated bilirubin levels earlier than 48 hours
* Discord with family

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of breast milk odor on phototherapy duration during phototherapy treatment. | Upon completion of the study, an average of 3 days
  While newborns received phototherapy treatment, cotton wool moistened with breast milk in a container was placed near the newborn's nose.
To evaluate the bilirubin level of breast milk odor during phototherapy treatment | Upon completion of the study, an average of 3 days
  While newborns received phototherapy treatment, cotton wool moistened with breast milk in a container was placed near the newborn's nose.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)